CLINICAL TRIAL: NCT04594135
Title: Anti-CD5 CAR T Cells for Relapsed/Refractory T Cell Malignancies
Acronym: CD5CAR-T
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: iCAR Bio Therapeutics Ltd. (Industry); Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICG190-001
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; T-cell Non-Hodgkin Lymphoma
Keywords: anti-CD5 CAR; T cell leukemia/lymphoma; T-ALL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell; Leukemia, T-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD5 CAR T cells (Experimental): Experimental: anti-CD5 CAR T cells Dose escalation phase: anti-CD5 CAR T cells transduced with a lentiviral vector to express CD5 chimeric receptor domain on T cells with an escalation approach, 1e6 to 5e6 CAR-T cells/kg
  Interventions: Drug: anti-CD5 CAR T cells

INTERVENTIONS:
Drug: anti-CD5 CAR T cells — anti-CD5 CAR T cells transduced with a lentiviral vector to express CD5 chimeric receptor domain on T cells

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of anti-CD5 CART cells in patients with relapsed and/or refractory T cell lymphoma or leukemia.

DETAILED DESCRIPTION:
Anti- CAR is a chimeric antigen receptor immunotherapy treatment designed to treat lymphoma/leukemia expressing CD5 antigen. CD5+ T cell lymphomas or leukemia are a subset of leukemias and lymphomas that are positive for the surface protein CD5. The purpose of this study is to evaluate the efficacy and safety of anti-CD5 CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent; Patients volunteer to participate in the research
2. Diagnosis is mainly based on the World Health Organization (WHO) 2008
3. Patients have exhausted standard therapeutic options
4. Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 1 weeks
5. Female must be not pregnant during the study

Exclusion Criteria:

1. Patients declining to consent for treatment
2. Prior solid organ transplantation
3. Potentially curative therapy including chemotherapy or hematopoietic cell transplant
4. Any drug used for GVHD must be stopped >1 week

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events after anti-CD5 CAR T cells cell infusion | 2 years particularly the first 28 days after infusion
  Determine the toxicity profile of anti-CD5 CAR T cell therapy

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | up to 6 months
  Incidence of treatment-emergent adverse events
Disease Free Survival (DFS) | up to 2 years
  Disease Free Survival (DFS)
Progression-Free Survival (PFS) | up to 2 years
  Progression-Free Survival (PFS)
Overall Survival (OS) | up to 2 years
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhang, MD/PhD, Principal Investigator — Peking University Shenzhen Hospital, China
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No